CLINICAL TRIAL: NCT00145353
Title: Is Insulin NovoRapid Better Than Actrapid for Treating Type 1 Diabetic Patients When Simultaneously, Daily Adjusting the Insulin Dose?
Brief Title: Insulin NovoRapid Versus Actrapid in Treatment of Type 1 Diabetic Patients During Daily Adjustment of Insulin Dose
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Odense University Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 007
Record Dates: First submitted 2005-09-02; First posted 2005-09-05 (Estimated); Last update posted 2006-10-11 (Estimated); Status verified 2006-10

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: type 1 diabetes mellitus; hypoglycaemia; insulin profiles; growth hormone; cortisol; glucagon
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia

INTERVENTIONS:
Drug: Insulin NovoRapid versus Actrapid

SUMMARY:
The main purpose of the study is to investigate the reason for the reduced number of hypoglycaemic attacks in type 1 diabetic patients when, for a period of time, using Insulin Aspart at meals together with NPH insulin mornings and evenings, and when, in another period of time, using human fast-working insulin at meals and NPH insulin mornings and evenings, and when the patients in both periods simultaneously take extra insulin at meals if high blood glucose values are found before meals.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus treated with insulin four times daily (basal bolus treatment) at least three months before screening.
* AGe: 18-60 years
* BMI: 18-27.5
* No nefro- or neuropathy; i.e. S-creatinin below 120 μmol/l and normal monofilament examination
* Written informed consent

Exclusion Criteria:

* Pregnant women or patients planning to become pregnant during the investigation period
* Reduced eyesight; i.e. visus > 0.3 evaluated at the latest eye exam.
* Patient lacking the ability to sens insulin sensitivity
* Serious rival disease, i.e. heart disease, severe liver or lung impairment, severe psychiatric disease.
* Suspicion of abuse or non-compliance
* Participation in another clinical trial

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16
Dates: Start 2004-11; Study Completion 2006-06

PRIMARY OUTCOMES:
Meal-regulated insulin time two peaks after the two intervention periods

CONTACTS AND LOCATIONS:
Overall Officials: Iben B. Jacobsen, MD, Principal Investigator — Odense University Hospital
Locations (1):
- Diabetes Research Center, Odense, Funen, Denmark